CLINICAL TRIAL: NCT01779700
Title: Safety and Efficacy of Fingolimod in Schizophrenia Patients Who Have Suboptimal Responses to Antipsychotic Drug Treatment
Brief Title: Fingolimod in Schizophrenia Patients
Acronym: STEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alan Breier, Psychiatrist, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11T-001
Record Dates: First submitted 2013-01-11; First posted 2013-01-30 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia
Keywords: psychosis; schizophrenia; cognition; fingolimod
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Fingolimod Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fingolimod (Active Comparator): 0.5mg of fingolimod, oral administration, daily, for 8 weeks.
  Interventions: Drug: Fingolimod
- placebo (Placebo Comparator): placebo, oral administration, daily, for 8 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fingolimod — 0.5mg each day of 8 week cycle
  Other Names: gilenya
  Arms: Fingolimod
Drug: placebo — 1 tablet each day of 8 week cycle
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
This will be a single site safety and proof of concept study conducted at the Indiana University Psychotic Disorders Program. Forty subjects with schizophrenia or schizoaffective disorders will be randomized 1:1 to double-blind treatment with fingolimod or matched placebo for duration of 8 weeks.

DETAILED DESCRIPTION:
Study Design:

This will be a single site safety and proof of concept study conducted at the Indiana University Psychotic Disorders Program. Forty subjects with schizophrenia or schizoaffective disorders will be randomized 1:1 to double-blind treatment with fingolimod or matched placebo for duration of 8 weeks.

All subjects will be admitted to the Indiana Clinical and Translational Sciences Institute Clinical Research Center (CRC) and remain hospitalized for the first 24 (+/- 2) hours post initial dose of study medication. The CRC is located in Indiana University Hospital and has 24 hour staffing with nurses skilled in conducting Phase 1 and Phase 2 investigational drug studies.

Background and Rationale:

Schizophrenia is a severe brain disorder that begins during the teenage years and early twenties and typically progresses to a life-long chronic illness marked by psychotic symptoms, cognitive impairment and poor functioning. A leading hypothesis to account for the symptoms and cognitive dysfunction of this disorder is that abnormalities exist in cortical circuits, particularly in frontal and temporal areas. An interest in cortical circuitry has led to a focus on the integrity of cortical white matter tracts as possibly contributing to the pathophysiology of this illness. Indeed, several lines of evidence have supported abnormalities in white matter structure and function in schizophrenia. Numerous myelin-related genes and their functional expression have been associated with schizophrenia. Moreover, quantitative and qualitative abnormalities in prefrontal cortical oligodendrocytes have been found in postmortem studies. MRI-determined volumetric reductions in prefrontal white matter have been reported in schizophrenia. Advances in MRI technology have enhanced the ability to study white matter pathology in vivo. Diffusion tensor imaging (DTI) and fractional anisotropy (FA) provides an assessment of the density and integrity of white matter tracts. Decreased FA has been reported in many de-myelinating diseases including multiple sclerosis (MS), leukodystrophies, and HIV. Numerous studies using DTI have reported decrements in FA in schizophrenia with the most consistent abnormalities occurring in frontal cortical white matter. Also, FA has been shown to be sensitive to therapeutic drug effects in MS which supports DTI-derived FA as an outcome measure in clinical trials of neuroprotective agents.

Fingolimod (FTY720, approved as Gilenya™ ) is a sphingosine-1-phosphate (S1P) receptor modulator and recently licensed in the USA and several other countries for relapsing forms of multiple sclerosis (MS). It is administered as a once per day oral preparation. In registration clinical trials, it had positive effects on brain atrophy, MRI-determined axonal lesions and relapse rates. Significant improvement in the mean number of MRI assessed T1 gadolinium (Gd) enhanced lesions/patient and the percentage of patients free of T1 Gd-enhanced lesions was observed within 6 months of treatment and there was evidence of clinical improvement as early as 2 months after treatment initiation

ELIGIBILITY:
Inclusion

* 18 to 65 yrs, able to give informed consent
* DSM IV-TR Diagnosis of schizophrenia or schizoaffective disorder
* Previous and/or current exposure to one of the following antipsychotic medications (clozapine, olanzapine, risperidone, paliperidone, haloperidol, quetiapine) as defined by a minimum of 8 weeks in duration greater than or equal to the Food and Drug Administration (FDA) approved therapeutic range for schizophrenia at the time of study entry OR previous and/or current exposure to two antipsychotic medications as defined by a minimum of 4 weeks in duration and greater than or equal to the FDA approved therapeutic range for schizophrenia at the time of study entry
* willing to participate in a minimum of 1 day of hospitalization
* Clinical stability:

  1. CGI-S score of < 4 at randomization AND
  2. no exacerbation of illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the investigator AND
  3. antipsychotic treatment stability for at least 4 weeks prior to randomization
* Female subjects of childbearing potential must test negative for pregnancy at screening and agree to use a single, effective, medically acceptable method of birth control for the duration of the study and for two months following cessation of study medication
* Subjects must agree not to consume tonic water for the duration of the study and for two months following cessation of study medication
* Sub-optimally treated positive OR negative symptoms as defined by the Brief Psychiatric Rating Scale (BPRS):

  1. BPRS positive symptom factor (conceptual disorganization, hallucinations, suspiciousness, unusual thought content) score of > 4 on any one item or a sum > 8 on the factor
  2. BPRS negative symptom factor (motor retardation, blunted affect, inappropriate affect) score of > 4 on any one item or a sum > 6 on the factor

Exclusion

* Subjects who are considered prisoners per the IU Standard Operating Procedures for Research Involving Human Subjects
* Current acute, serious, or unstable medical conditions
* Clinically significant electrocardiogram abnormality: corrected QT interval >450 msec (M) or >470 msec (F) prior to randomization OR sinus bradycardia (HR < 50 beats/min)
* Subjects who have experienced the following within the six months prior to study entry: myocardial infarction, unstable angina, stroke, transient ischemic attach (TIA), decompensated heart failure requiring hospitalization or Class III/IV heart failure
* Hypokalemia, hypomagnesemia, or congenital long-QT syndrome
* Known HIV+ status
* Active seizure disorder
* Pregnant or lactating women or women who plan to become pregnant or will be lactating within two months after cessation of study drug
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, ventriculoperitoneal shunt, or other contraindication to undergoing an MRI scan
* Class1a or class 3 antiarrhythmic agents, beta blockers, diltiazem, verapamil, digoxin, tricyclic antidepressants, warfarin, ketoconazole, ketamine
* Subjects likely to need a live attenuated vaccine during the course of the study or within two months after stopping study medication
* Subjects with no history of chicken pox or chicken pox vaccination, or with a negative VZV titer
* Active herpes simplex outbreak, mononucleosis, or zoster
* Subjects with histories of ischemic heart disease, myocardial infarction, congestive heart failure, cardiac arrest, cerebrovascular disease, unexplained or recurrent syncope, cardiac conduction prolongations (prolonged P-R interval), cardiac arrhythmias, symptomatic bradycardia, or severe untreated sleep apnea
* Antineoplastic, immunosuppressive, or immune modulating therapies
* History of macular edema or uveitis
* Known IQ < 70
* Current active fungal or viral infection
* Current DSM IV-TR diagnosis of substance dependence (excluding caffeine and nicotine)
* Positive urine toxicology screen for the following: cocaine, barbiturates, methamphetamine, opiate, methadone, phencyclidine, or amphetamine prior to randomization
* Test positive for (1) Hep C virus antibody, (2) Hep B surface antigen (HBsAg) with or without positive Hep B core total antibody, (3) HIV 1 or 2 antibodies, or (4) Mantoux tuberculin test.
* Moderate to severe renal impairment as defined by creatinine clearance < 60 ml/min at screening
* Hepatic impairment as defined by liver transaminases or total bilirubin > 3 × upper limit of normal
* Subjects considered a high risk for suicidal acts - active suicidal ideation OR any suicide attempt in 90 days prior to screening
* Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to screening OR Subjects currently receiving treatment (within 1 dosing interval + 4 weeks) with an investigational depot formulation of an antipsychotic medication
* Subjects who demonstrate overtly aggressive behavior or who are deemed to pose a homicidal risk in the investigator's opinion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Breier, MD, Principal Investigator — Indiana University; Michael Francis, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Center for NeuroImaging, Indianapolis, Indiana
  - Prevention and Recovery Center, Indianapolis, Indiana
  - Larue D Carter Memorial Hospital, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fingolimod | Placebo
Started | 18 | 22
Completed | 14 | 17
Not Completed | 4 | 5
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 22 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.33 (10.28) | 37.00 (13.19) | 36.70 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 8 | 8 | 16
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: QTcB Change
Description: To determine the safety of fingolimod, as measured by the electrocardiogram (ECG) QT interval corrected by Bazett's (QTcB) value.
Time Frame: Screening, Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 84, Day 112
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
ms
  QTcB - Screening | 416.50 (19.24) | 416.41 (17.69)
  QTcB - Day 0 | 418.39 (23.47) | 423.27 (22.05)
  QTcB - Day 7 | 415.50 (16.71) | 417.00 (19.99)
  QTcB - Day 14 | 418.28 (16.30) | 420.15 (16.24)
  QTcB - Day 21 | 419.67 (18.90) | 412.00 (19.25)
  QTcB - Day 28 | 424.06 (17.51) | 415.74 (18.26)
  QTcB - Day 35 | 426.18 (25.31) | 419.00 (20.47)
  QTcB - Day 42 | 425.53 (22.10) | 414.33 (17.81)
  QTcB - Day 49 | 420.79 (24.50) | 413.53 (18.02)
  QTcB - Day 56 | 420.67 (21.25) | 418.41 (18.38)
  QTcB - Day 84 | 421.50 (26.18) | 420.68 (22.69)
  QTcB - Day 112 | 419.67 (20.22) | 418.58 (18.88)

2. Primary Outcome: Levels of Lymphocyte
Description: To determine the safety of fingolimod, as measured by the absolute lymphocyte count
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: 10^3 lymphocytes/uL
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
10^3 lymphocytes/uL
  Absolute lymphocyte count - Baseline | 1.99 (0.57) | 1.97 (0.64)
  Absolute lymphocyte count - 4 weeks | 0.44 (0.22) | 1.94 (0.47)
  Absolute lymphocyte count - 8 weeks | 0.49 (0.32) | 2.00 (0.76)

3. Primary Outcome: Symptom Changes - PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a semi-structured interview, containing 30 items that assess symptoms of psychotic disorders including positive, negative, and general psychopathology symptoms. Positive symptoms are rated on 7 items, negative symptoms are rated on 7 items, and general psychopathology on 16 items. Scores for each item range from 1=absent to 7=extreme. Positive, negative, and general psychopathology symptoms can each respectively render total scores. Positive total scores ranging from 7-49, negative total scores ranging from 7-49, and general psychopathology scores ranging from 16-112. When all items are summed together a total score is generated. Total scores for all items range from 30-210, a lower score reflecting fewer symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale
  PANSS Total Score - Baseline | 48.89 (11.58) | 56.50 (11.17)
  PANSS Total Score - 4 weeks | 49.78 (14.69) | 53.60 (12.17)
  PANSS Total Score - 8 weeks | 49.06 (14.65) | 54.94 (11.53)

4. Secondary Outcome: Verbal Memory - BACS
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is a battery specifically designed to measure treatment-related changes in cognition. The BACS utilizes 6 tasks, and has alternate forms, thus minimizing practice effects. Each task generates a raw score (with a higher score indicating better performance): verbal memory 0-75; digit sequencing 0-28; token motor task 0-100; semantic&letter fluency 0-148; symbol coding 0-110; and tower of London 0-22. The raw scores are used to generate a composite score that is calculated by summing t-scores derived by comparisons with a normative sample of 404 healthy controls. The six brief assessments' t-scores, are summed, and averaged to provide a composite t-score. The composite score min and max are between -43 and 100. A higher score indicating better cognitive performance.
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale
  BACS Verbal Memory - Baseline | 30.89 (9.61) | 37.45 (11.65)
  BACS Verbal Memory - 4 weeks | 33.50 (8.87) | 35.45 (9.56)
  BACS Verbal Memory - 8 weeks | 34.69 (10.62) | 36.11 (11.53)

5. Secondary Outcome: Cognition Change - BACS
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is a battery specifically designed to measure treatment-related changes in cognition by utilizing 6 tasks, and has alternate forms, thus minimizing practice effects. Each task generates a raw score (with a higher score indicating better performance): verbal memory 0-75; digit sequencing 0-28; token motor task 0-100; semantic&letter fluency 0-148; symbol coding 0-110; and tower of London 0-22. The raw scores are used to generate a composite score that is calculated by summing t-scores derived by comparisons with a normative sample of 404 healthy controls. The six brief assessments' t-scores, are summed, and averaged to provide a composite t-score. The composite score min and max are between -43 and 100. A higher score indicating better cognitive performance.
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale
  BACS Composite Score - Baseline | 25.17 (14.75) | 30.95 (9.48)
  BACS Composite Score - 4 weeks | 27.67 (13.61) | 32.10 (10.64)
  BACS Composite Score - 8 weeks | 31.13 (12.52) | 33.50 (11.45)

6. Secondary Outcome: Cognition Change - Trails B
Description: The Trail Making Test-Part B (Trails B) is a measure of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive targets on a sheet of paper. In Part B version the subject alternates between numbers and letters (1, A, 2, B, etc.) The goal of the test is for the subject is to finish part B as quickly as possible, the time taken to complete the test is used as the primary performance metric. The score is the number of seconds it took to complete the test.
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
seconds
  Trails B - Baseline | 108.00 (51.86) | 123.64 (71.11)
  Trails B - 4 weeks | 97.88 (40.57) | 100.60 (48.02)
  Trails B - 8 weeks | 84.53 (28.79) | 102.33 (74.48)

7. Secondary Outcome: Positive Symptom Change - PANSS
Description: as for outcome 3
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale
  PANSS Positive Score - Baseline | 10.83 (4.94) | 13.64 (5.59)
  PANSS Positive Score - 4 weeks | 11.89 (6.24) | 14.00 (5.52)
  PANSS Positive Score - 8 weeks | 10.06 (4.74) | 13.06 (5.40)

8. Secondary Outcome: Negative Symptom Change - PANSS
Description: as for outcome 3
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale
  PANSS Negative Score - Baseline | 15.00 (4.79) | 16.59 (5.32)
  PANSS Negative Score - 4 weeks | 13.89 (3.53) | 14.80 (5.20)
  PANSS Negative Score - 8 weeks | 15.44 (4.35) | 15.06 (4.67)

9. Secondary Outcome: Plasma Cytokines Levels - IL-10
Description: To assess IL-10 plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL10 - Baseline | 16.11 (20.81) | 11.94 (13.38)
  IL10 - 4 weeks | 15.50 (20.67) | 9.23 (10.68)
  IL10 - 8 weeks | 16.28 (20.96) | 10.42 (9.84)

10. Secondary Outcome: Plasma Cytokines Levels - IL-17A
Description: To assess IL-17A plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL17A - Baseline | 3.09 (3.03) | 3.72 (6.87)
  IL17A - 4 weeks | 2.58 (2.39) | 2.43 (2.15)
  IL17A - 8 weeks | 2.58 (2.36) | 2.69 (2.27)

11. Secondary Outcome: Plasma Cytokines Levels - IL-1BETA
Description: To assess IL-1BETA plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL1BETA - Baseline | 0.87 (0.81) | 0.69 (0.53)
  IL1BETA - 4 weeks | 0.81 (0.82) | 0.72 (0.63)
  IL1BETA - 8 weeks | 0.82 (0.76) | 0.74 (0.68)

12. Secondary Outcome: Plasma Cytokines Levels - IL-2
Description: To assess IL-2 plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL2 - Baseline | 1.74 (2.42) | 1.27 (1.43)
  IL2 - 4 weeks | 1.96 (2.95) | 1.20 (1.63)
  IL2 - 8 weeks | 1.77 (2.55) | 1.20 (1.24)

13. Secondary Outcome: Plasma Cytokines Levels - IL-4
Description: To assess IL-4 plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL4 - Baseline | 30.99 (30.86) | 30.74 (33.76)
  IL4 - 4 weeks | 27.40 (23.61) | 31.34 (31.24)
  IL4 - 8 weeks | 24.20 (24.57) | 32.16 (34.78)

14. Secondary Outcome: Plasma Cytokines Levels - IL-6
Description: To assess IL-6 plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL6 - Baseline | 2.15 (2.28) | 1.90 (1.75)
  IL6 - 4 weeks | 2.22 (2.62) | 1.81 (1.99)
  IL6 - 8 weeks | 2.16 (2.66) | 1.96 (1.56)

15. Secondary Outcome: Plasma Cytokines Levels - IL-8
Description: To assess IL-8 plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IL8 - Baseline | 4.29 (5.55) | 3.83 (4.63)
  IL8 - 4 weeks | 3.81 (3.71) | 3.69 (4.28)
  IL8 - 8 weeks | 4.18 (4.77) | 3.69 (4.00)

16. Secondary Outcome: Plasma Cytokines Levels - TNFa
Description: To assess TNFa plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  TNFa - Baseline | 2.11 (2.16) | 1.76 (1.32)
  TNFa - 4 weeks | 2.02 (2.77) | 1.86 (1.38)
  TNFa - 8 weeks | 2.00 (2.19) | 1.61 (1.09)

17. Secondary Outcome: Plasma Cytokines Levels - IFNgamma
Description: To assess IFNgamma plasma cytokines levels changes in participants taking fingolimod versus placebo
Time Frame: Baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 18 | 22
pg/ml
  IFNgamma - Baseline | 5.32 (4.17) | 8.32 (16.21)
  IFNgamma - 4 weeks | 4.61 (3.54) | 4.95 (3.70)
  IFNgamma - 8 weeks | 4.32 (3.38) | 5.62 (4.40)

ADVERSE EVENTS:
Time Frame: Screening through day 112
Arm/Group | Fingolimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/22
Other Adverse Events (participants affected / at risk) | 18/18 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingolimod (N=18) | Placebo (N=22)
Hospitalization for exacerbation of schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingolimod (N=18) | Placebo (N=22)
Asymptomatic Bradycardia (Cardiac disorders) | 3 (3) | 3 (4)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
headache (General disorders) | 3 (3) | 2 (2)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
QTc Interval Prolongation (Cardiac disorders) | 2 (2) | 0 (0)
Mobitz I AV Block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension, intermittent (Cardiac disorders) | 1 (1) | 0 (0)
Lymphocytopenia (Blood and lymphatic system disorders) | 18 (18) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 5 (5) | 0 (0)
Blurry vision (Eye disorders) | 3 (3) | 0 (0)
Dry mouth (General disorders) | 2 (2) | 0 (0)
Exacerbation of Allergic Rhinitis (General disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
mood lability (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Increased auditory hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Paresthesia (General disorders) | 1 (1) | 1 (1)
Stuttering (General disorders) | 1 (1) | 0 (0)
Dyskinetic Movement (General disorders) | 1 (1) | 0 (0)
Worsening of intermittent panic attacks (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT01779700/Prot_SAP_000.pdf